CLINICAL TRIAL: NCT06062615
Title: Randomized Pilot Study Investigating Early Functional Outcomes With the Use of Robotic Assisted Versus Conventional Total Knee Arthroplasty"
Brief Title: Robotic Assisted TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAUS 22D.103
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Total knee replacement (TKR) without Omnibot system (Active Comparator): The participant will undergo TKR utilizing conventional techniques.
  Interventions: Procedure: Conventional Total knee replacement
- Total knee replacement (TKR) with Omnibot (Active Comparator): The participant will undergo a robotic assisted TKR utilizing the Omnibot Knee System
  Interventions: Procedure: Total knee replacement using Omnibot Knee System; Device: Omnibot Robotic Knee System

INTERVENTIONS:
Procedure: Total knee replacement using Omnibot Knee System — total knee replacement with robotic assistance
  Arms: Total knee replacement (TKR) with Omnibot
Procedure: Conventional Total knee replacement — Conventional total knee replacement without robotic assistance
  Arms: Total knee replacement (TKR) without Omnibot system
Device: Omnibot Robotic Knee System — utilizes an active motorized knee spacer to measure ligament tension and gap balance after the tibia has been cut during surgery
  Arms: Total knee replacement (TKR) with Omnibot

SUMMARY:
As an intraoperative tool, a modern robotic total knee arthroplasty (TKA) system should be able to identify a patient's native femoral and tibial anatomy, as well as, assess ligament tension and gap balance. The surgeon in real time is then able to develop and execute a patient specific plan in terms of component size, alignment and rotation. In our institution we have begun to use, the OMNIBotics Knee system (Corin), which utilizes an active motorized knee spacer, BalanceBot, to objectively measure ligament tension and gap balance after the tibia has been cut and its alignment confirmed. This information is then processed through the OMNIbotics computer algorithm to appropriately size, align, and rotate the femur component to balance the flexion and extension gaps. The purpose of this study is to perform a randomized pilot study looking for an effect on early functional outcomes comparing robotic assisted TKA (RATKA) versus conventional TKA technique.

ELIGIBILITY:
Inclusion Criteria:

* All unilateral primary knee arthroplasties performed by the investigator participating in this study will be eligible for inclusion
* Diagnosis of primary osteoarthritis

Exclusion Criteria:

* Revision surgery
* Bilateral knee surgery
* Age <18 or >80
* BMI >40
* Baseline lower extremity strength less than 5/5
* History of chronic narcotic use, defined as more than 5mg of oxycodone q4 hours
* Functionally limiting spine disease
* Other functionally limiting lower extremity disorder (i.e. symptomatic ipsilateral hip disease)
* Patients who cannot perform the baseline functional tests
* Allergy/contraindication to protocol medications
* Post-traumatic arthritis
* Inflammatory arthritis
* Pregnancy
* Prisoners
* Patients receiving care as a result of a worker's compensable injury
* General anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
early functional outcomes #1 | 6 months
  This will be measured by the timed-up-and-go test.
Early functional outcomes #2 | 6 months
  This will be measured by the stair climbing test.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Austin, MD, Principal Investigator — Rothman Orthopaedic Institute
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lizcano JD, Restrepo S, Tarabichi S, Gold PA, Saxena A, Austin MS. Does the Use of a Robotic Gap-tensioning System Improve Functional Outcomes After TKA? A Randomized Clinical Trial. Clin Orthop Relat Res. 2025 Oct 22. doi: 10.1097/CORR.0000000000003734. Online ahead of print. PMID 41191410